CLINICAL TRIAL: NCT01485250
Title: A Cross-Cultural Assessment of the Motivations of Healthy Participants in Phase I Research
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 999910061; 10-CC-N061
Record Dates: First submitted 2011-11-30; First posted 2011-12-05 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-08-08

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteers; Motivations; Decision Making; Motivation

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Individuals often participate in clinical trials to seek new therapies and free medical treatments for their illnesses or chronic conditions. However, less is known about the motivations of the healthy individuals who volunteer for research studies.
* Although many healthy volunteers participate in clinical trials for financial compensation, the particular risks involved in testing drugs that have not been tried in human clinical trials pose potential dangers for healthy volunteers in Phase I studies. More research is needed to understand the motivations of volunteers who participate in Phase I clinical trials.

Objectives:

- To evaluate the primary and secondary motivations of healthy participants in research studies.

Eligibility:

- Individuals at least 18 years of age who are healthy volunteers in selected Pfizer Phase I clinical trials.

Design:

* Individuals who express interest in participating in specific Pfizer Phase I drug studies will be asked to complete a short questionnaire after completing the standard consent session for the study.
* Those who enroll in the trial will be asked to complete a second questionnaire prior to discharge from the study.

DETAILED DESCRIPTION:
This healthy volunteer motivation study is a sub-study of Phase I drug development studies conducted by Pfizer International. The substudy is designed to evaluate the primary and secondary motivations of healthy participants in research studies, as well as the process by which participants decide to participate, including their consideration of any risks, benefits, compensation and other factors, and the relationship of these factors to cultural and sociodemographic variables. Data will be collected via self-administered surveys at 2 possible time points, 1) after going through the consent process at the beginning of participation in the primary study, and 2) towards the end of the study participation.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be willing adults who have participated in an informed consent session for a designated Phase I study at a Pfizer CRU. Participants in New Haven and Singapore must be able to read and answer question in English and participants in Brussels must be able to read and answer questions either in English, French, or Flemish. Only adults (over 18 years old) who can provide their own consent will be included.

EXCLUSION CRITERIA:

Participants in Pfizer phase I studies who are unable or unwilling to complete the survey instruments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1278 (Actual)
Dates: Start 2010-02-19; Study Completion 2018-08-08

CONTACTS AND LOCATIONS:
Overall Officials: Christine Grady, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (3):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Pfizer CRU, Brussels, Belgium
- Pfizer CRU, Singapore, Singapore

REFERENCES:
- [Background] Almeida L, Azevedo B, Nunes T, Vaz-da-Silva M, Soares-da-Silva P. Why healthy subjects volunteer for phase I studies and how they perceive their participation? Eur J Clin Pharmacol. 2007 Nov;63(11):1085-94. doi: 10.1007/s00228-007-0368-3. Epub 2007 Sep 20. PMID 17891536
- [Background] Bigorra J, Banos JE. Weight of financial reward in the decision by medical students and experienced healthy volunteers to participate in clinical trials. Eur J Clin Pharmacol. 1990;38(5):443-6. doi: 10.1007/BF02336681. PMID 2379528
- [Background] Cunny KA, Miller HW. Participation in clinical drug studies: motivations and barriers. Clin Ther. 1994 Mar-Apr;16(2):273-82; discussion 271-2. PMID 8062322